CLINICAL TRIAL: NCT03666676
Title: Auditory Processing of Complex Sounds - Sensitivity to Chirps
Brief Title: Hearing Study: Sensitivity to Features of Speech Sounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Laurel Carney, Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 73346; R01DC001641 (NIH)
Record Dates: First submitted 2018-09-08; First posted 2018-09-12 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Hearing (Active Comparator): Signal processing to improve intelligibility
  Interventions: Other: Signal processing to improve intelligibility
- Mild hearing loss (Active Comparator): Signal processing to improve intelligibility
  Interventions: Other: Signal processing to improve intelligibility
- Moderate hearing loss (Active Comparator): Signal processing to improve intelligibility
  Interventions: Other: Signal processing to improve intelligibility

INTERVENTIONS:
Other: Signal processing to improve intelligibility — Signal processing will be used to manipulate frequency and amplitude fluctuations in complex sounds.

SUMMARY:
The purpose of this study is to better understand the sensitivity of listeners to the fast changes in frequency or amplitude of sounds that occur in speech. The investigators are studying ways to manipulate these aspects of sounds in an effort to make speech sounds more clear.

DETAILED DESCRIPTION:
The investigators will test listeners with normal hearing or with mild or moderate hearing loss. Tests will first focus on sensitivity to changes in fast changes in amplitude (loudness) or frequency (pitch) in sounds. Then the investigators will test the intelligibility of synthetic vowels and syllables in which these "chirps" are manipulated. Finally, the investigators will test intelligibility of words in noise while manipulating sounds in an effort to improve clarity.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing, mild or moderate symmetric sensorineural hearing loss.

Exclusion Criteria:

* Asymmetric hearing thresholds (more than 15 decibels (dB) threshold difference between the two ears at any frequency up to 4 kHz).
* Severe hearing loss (greater than 60 dB hearing thresholds at any frequency up to 4 kHz).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel H Carney, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carney LH, Cameron DA, Kinast KB, Feld CE, Schwarz DM, Leong UC, McDonough JM. Effects of sensorineural hearing loss on formant-frequency discrimination: Measurements and models. Hear Res. 2023 Aug;435:108788. doi: 10.1016/j.heares.2023.108788. Epub 2023 May 8. PMID 37224720

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Hearing | Mild Hearing Loss | Moderate Hearing Loss
Started | 36 | 16 | 15
Completed | 23 | 8 | 3
Not Completed | 13 | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hearing | Mild Hearing Loss | Moderate Hearing Loss | Total
Number analyzed (Participants) | 36 | 16 | 15 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 7 | 6 | 48
  >=65 years | 1 | 9 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (15) | 60 (11) | 60 (19) | 45 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 9 | 42
  Male | 16 | 3 | 6 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 1 | 5
  Not Hispanic or Latino | 32 | 16 | 14 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 1 | 0 | 7
  White | 26 | 14 | 15 | 55
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 16 | 15 | 67
Audiometric Thresholds [Mean (Standard Deviation); unit: decibels] — Audiometric thresholds of subjects at 2000 Hz, a frequency where formant-frequency discrimination was measured.
  decibels | 5.5 (7.0) | 23.8 (5.2) | 46.1 (6.9) | 17.0 (17.7)

OUTCOME MEASURES:

1. Primary Outcome: Pure-tone Average Thresholds
Description: Hearing thresholds, average across test frequencies from 250 to 4000 Hz and averaged across the two ears.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Hearing level in dB SPL
Groups:
- Normal Hearing: Participants with normal hearing
- Mild Hearing Loss: Participants with mild hearing loss
- Moderate Hearing Loss: Participants with moderate hearing loss.
Arm/Group | Normal Hearing | Mild Hearing Loss | Moderate Hearing Loss
Number analyzed (Participants) | 23 | 8 | 3
Hearing level in dB SPL | 7.3 (6.3) | 30.8 (6.0) | 46.9 (6.6)

2. Primary Outcome: F1 Discrimination Threshold
Description: Discrimination threshold for changes in F1, the low-frequency formant (spectral peak) in the synthetic vowel sounds.
Time Frame: 6 months
Population: The analysis populations were determined based on the pure-tone average thresholds (outcome measure 1)
Measure: Mean (Standard Deviation); unit: % frequency
Groups:
- Normal Hearing: Participants with a normal hearing
Arm/Group | Normal Hearing | Mild Hearing Loss | Moderate Hearing Loss
Number analyzed (Participants) | 23 | 8 | 3
% frequency | 5 (2.3) | 7.8 (5.5) | 5.9 (2.0)

3. Primary Outcome: F2 Discrimination Threshold
Description: Discrimination thresholds in % frequency for F2, the higher-frequency peak in synthetic vowel stimuli.
Time Frame: 6 month
Population: The groups of subjects were determined by the pure tone average thresholds, from Outcome Measure 1.
Measure: Mean (Standard Deviation); unit: % frequency
Groups:
- Normal Hearing: Listeners with normal hearing
- Mild Hearing Loss: Listeners with mild hearing loss
- Moderate Hearing Loss: Listeners with moderate hearing loss
Arm/Group | Normal Hearing | Mild Hearing Loss | Moderate Hearing Loss
Number analyzed (Participants) | 23 | 8 | 3
% frequency | 4 (2.9) | 21 (11.3) | 30.8 (6.2)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Normal Hearing; Mild Hearing Loss; Moderate Hearing Loss: Signal processing to improve intelligibility
  Signal processing to improve intelligibility: Signal processing will be used to manipulate frequency and amplitude fluctuations in complex sounds.
  No Adverse events occurred.
Arm/Group | Normal Hearing | Mild Hearing Loss | Moderate Hearing Loss
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/36 | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03666676/Prot_SAP_000.pdf